CLINICAL TRIAL: NCT04366167
Title: An Observational Cohort Study to Explore Patient Outcome From Heart Surgery During the Covid-19 Pandemic (CardiacCovid)
Brief Title: Patient Recovery From Heart Surgery During the Covid-19 Pandemic
Acronym: CardiacCovid
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 132127
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2021-10

CONDITIONS: Cardiac Surgery; COVID
Keywords: cardiac surgery; patient reported outcomes; COVID
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cardiac surgery patients - lockdown 1: Cohort 1 (lockdown 1): Patients undergoing adult cardiac surgery during the Covid-19 pandemic
  Interventions: Other: Cardiac surgery
- Cardiac surgery patients - lockdown 2: Cohort 2 (lockdown 2): Patients undergoing adult cardiac surgery during the Covid-19 pandemic
  Interventions: Other: Cardiac surgery
- Cardiac surgery patients - lockdown 3: Cohort 3 (lockdown 3): Patients undergoing adult cardiac surgery during the Covid-19 pandemic
  Interventions: Other: Cardiac surgery

INTERVENTIONS:
Other: Cardiac surgery — Cardiac surgery during the COVID-19 pandemic

SUMMARY:
This study will describe and explore the recovery process of patients undergoing cardiac surgery during the covid-19 pandemic. This will include mortality, morbidity, health-related quality of life, event-specific distress and depression.

DETAILED DESCRIPTION:
The overall aim of this study is to describe and explore the recovery process of patients undergoing cardiac surgery during the covid-19 pandemic. This will include mortality, morbidity, health-related quality of life, event-specific distress and depression.

All adult patients having cardiac surgery during the pandemic at St Bartholomew's Hospital will be approached to join this study. As of the end of March this is this is approximately 20 operations a week. Questionnaires will be administered at five time points alongside a review of clinical notes.

Appropriate descriptive and summative statistics will be used to analyse outcomes. If sample size is adequate, possible associations/effect of the impact of the covid-19 pandemic on each of the recovery parameters included in the study will be determined. The differences in outcomes between those with and without covid-19 may also be analysed if the sample size is adequate. Bias and loss to follow-up in observational cohort studies has been considered.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiac surgery during the Covid-19 pandemic (end date as yet unknown but inferred when elective surgery is reinstated)
* Discharge from hospital where operation was performed is being planned
* Able and willing to give informed consent

Exclusion Criteria:

* Unable or unwilling to give written informed consent. This includes patients who are being transferred to another hospital and are considered too vulnerable or unwell to be approached (based on clinical judgement of the clinical care team)
* Unable or unwilling to give and/or complete the questionnaires
* Inability to understand written and/or verbal English

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery during the COVID-19 pandemic
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2020-04-18 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Change in Impact of Events scores | Baseline, 1 week after discharge, 6 weeks (+/- 2 weeks) post surgery, 6 months (+/- 2 weeks) post surgery, 1 year (+/- 2 weeks) post surgery
  The revised Impact of Events revised version (IES-R) questionnaire (Weiss and Marmar, 1997) is widely used as a measure of event-specific distress and measures distress experienced by serious life changes/events. It has been commonly used to assess persons with posttraumatic stress disorder (PTSD). It is an 22 item self-report scale where is item is reported on a five point likert scale from 0 (not at all) to 4 (extremely) with respect to how distressing each item has been during the past week. Scale scores are formed for the three subscales, which reflect intrusion (8 items: 1, 2, 3, 6, 9, 14, 16, 20), avoidance (8 items: 5,7,8,11,12,13,17,22), and hyperarousal (6 items: 4,10,15.18.19.21). A cut-off of 26 and above has been suggested for a clinically significant reaction to a psychological trauma, although the IES alone does not diagnose PTSD or reflect a person's ability to function. Metric for summarising data: t-test

SECONDARY OUTCOMES:
Survival | Up to 1 year post surgery
  Death or survival after cardiac surgery
Morbidity | Up to 1 year post surgery
  patient completion of a log sheet documenting all 'visits' (including calls to NHS 111, face-to-face or virtual visits) to the emergency department, hospital admissions and visits to the general practitioner on a standardised proforma for the duration of the study
Change in Health-related quality of life scores | Baseline, 1 week after discharge, 6 weeks (+/- 2 weeks) post surgery, 6 months (+/- 2 weeks) post surgery, 1 year (+/- 2 weeks) post surgery
  Health-related quality of life will be measured using the EQ5D-5L questionnaire. The EQ5D is a standardised, simple generic measure of health well, which is received by patients (Kim et al., 2005). It consists of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each with five levels of health response and a visual analogue scale (VAS) ranging from 0-100 (0 being the worst possible health imaginable and 100 being the best possible health imaginable). Metric for summarising data: t-test
Change in Depression scores | Baseline, 1 week after discharge, 6 weeks (+/- 2 weeks) post surgery, 6 months (+/- 2 weeks) post surgery, 1 year (+/- 2 weeks) post surgery
  Depression will be measured using the Centre for Epidemiologic Studies Depression Scale (CES-D). The CES-D is a 20-item self-report adult instrument designed to measure common symptoms of depression that have occurred over the past week, such as poor appetite, hopelessness, pessimism, and fatigue. All questions are answered on a scale of 0-3, with 0 indicating no symptom presence and with 3 representing symptoms "most or all of the time." CES-D scores range from 0 to 60 with higher scores indicating more severe depressive symptoms. A score of 16 or higher identifies subjects with clinically meaningful depression. Metric for summarising data: t-test

CONTACTS AND LOCATIONS:
Overall Officials: Julie Sanders, PhD, Principal Investigator — St. Bartholomew's Hospital
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Sanders J, Beaumont E, Dodd M, Murray SE, Owens G, Berry A, Hyde E, Bueser T, Clayton T, Oo AY. The impact of the COVID-19 pandemic on recovery from cardiac surgery over time: results of the CardiacCovid study from three UK national lockdowns. Eur J Cardiovasc Nurs. 2024 May 28;23(4):418-422. doi: 10.1093/eurjcn/zvad084. PMID 37585652
- [Derived] Sanders J, Bueser T, Beaumont E, Dodd M, Murray SE, Owens G, Berry A, Hyde E, Clayton T, Oo AY. The impact of the COVID-19 pandemic on recovery from cardiac surgery: 1-year outcomes. Eur J Cardiovasc Nurs. 2023 Jul 19;22(5):516-528. doi: 10.1093/eurjcn/zvac083. PMID 36099505